CLINICAL TRIAL: NCT01568801
Title: Evaluation of the Singapura Program of All Inclusive Care for the Elderly
Brief Title: Evaluation of the Singapura Program of All Inclusive Care for the Elderly (SingaPACE) Demonstration Project
Acronym: SingaPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Singapore General Hospital (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Dr. David Matchar, Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2011/381/A; 2011/381/A (Other: Singapore Health CIRB)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Frail Elders
Keywords: Integrated Services; Health Services for the Elderly; Community Services

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Individuals randomized into the control arm will receive usual community care services referred by the social worker from SGH and AH.
- Intervention Group (Experimental): Individuals in the intervention group will go through an integrated program of community based health and social care based on intake and ongoing evaluation by the SingaPACE team.
  Interventions: Behavioral: SingaPACE

INTERVENTIONS:
Behavioral: SingaPACE — Individuals in the intervention group will go through an integrated program of community based health and social care, based on intake and ongoing evaluation by the SingaPACE team.
  Arms: Intervention Group

SUMMARY:
This is a RCT studying the effectiveness of the Singapore Program for All Inclusive Care for the Elderly (SingaPACE) demonstration project over a 36 month period. SingaPACE is modelled on the US PACE home and community based service that acts as an alternative to institutional care. The comparator is best referrals for care as currently arranged through the Agency for Integrated Care (AIC) and referred by medical social workers. This research aims to determine how the SingaPACE model of health and social care affects use of emergency and acute care hospital services, institutional care, the quality of life (QOL) and satisfaction of the participants aged 60+ and their caregivers.

The hypotheses to be tested are:

H01: The elderly in SingaPACE will have fewer admissions to accident & emergency (A&E) hospitalization than the elderly who are not in SingaPACE.

H02: The elderly in SingaPACE will have fewer admissions to acute care hospitalization than the elderly who are not in SingaPACE.

H03: The elderly in SingaPACE will delay first admission to institutionalized nursing home care more than the elderly who are not in SingaPACE.

H04: The elderly in SingaPACE clients will have a higher QOL compared to the elderly who are not in SingaPACE.

H05: Caregivers of the elderly in SingaPACE will have a lower care-giving burden compared to caregivers of the elderly who are not in SingaPACE.

DETAILED DESCRIPTION:
* Recruitment

Potential subjects will be identified from i) inpatients referred prior to discharge and ii) outpatients to medical social workers from Singapore General Hospital (SGH) and Alexandra Hospital (AH). After confirming study eligibility the medical social worker will inform the potential subject about the study; after obtaining informed consent, the medical social worker will make a telephone call to the Duke - NUS research fellow who will then carry out the randomization process, assigning the subject to either the intervention group or the control group.

* Sites

The SingaPACE program will be located at 298, Tiong Bahru Road, #15-01/06 Central Plaza and at NTUC Eldercare, Block 117, Bukit Merah View.

* Procedures

* Randomization will be stratified at each recruitment site by gender, assuring equal numbers of men and women in each study arm; and by hospital assuring equal number of patients from SGH and AH in each study arm. 20 participants will enter the study (10 per arm) each month over a proposed 4-month recruitment period. If the recruitment rate is lower than expected, the recruitment period will be extended.
* Individuals in the intervention group will have a program of services based on intake and ongoing evaluation using interRAI by the SingaPACE assessment team. Services included in the integrated available mix are:

  * Case management across the continuum of care
  * Medical care by the SingaPACE physician
  * Home nursing (e.g., for administering parenteral medication, wound care, assessment of health status, nutrition)
  * Home care (e.g., for assistance with ADL)
  * Physiotherapy
  * Occupational therapy
  * Psychosocial care and counseling by social workers
  * Transportation to care and support services
  * Emergency housing and beds - public hospital acute bed substitution

    24 hour doctor / nurse phone coverageIf individuals in the intervention group leave the SingaPACE program, they will still continue to be tracked as a part of intention-to-treat analysis. Patients who die over the 36 months will be counted as drop outs. While the program can have new replacements for patients who have died, new participants will not be counted as a part of the intervention group in this research study.
* Individuals randomized to the control arm will be referred to the medical social worker for referral to community services as usual. The control group will be interviewed on their medical history, healthcare utilization and expenditure data. The data collected will be complemented by data that may be made available by the VWO providing home and community care to the control group. Such VWO data may possibly include assessments using RAF.

If participants from the control group switch from a VWO community care program to another VWO community care program, they will still continue to be tracked and included in the intention-to-treat analysis. For participants who die over the period of study, they will be counted as loss to follow-up.

The control group will receive community care services referred by the SGH MSW:

* VWO community care
* GPs
* Polyclinics
* Specialist Outpatient Clinics
* Traditional Chinese Medicine or herbal treatments
* Supportive care arrangements of the family, relatives and friends

  * All participants will be tracked over a 36-month period starting August 2011. Following the US PACE impact evaluation from 1998 observations of all patients will be made at the beginning of the intervention and follow up at 6 month intervals (Chatterji et al. 1998; Irvin, Massey and Dorsey 1997; White, Abel and Kidder, 2000).

Analysis The main outcome measure is number of EMT events, A&E events and acute care events over the 36 month period. This is the primary endpoint.

The secondary endpoints to be studied are time to first admission to nursing home over the 36 month period, LOS in A&E; LOS in acute care; patient QOL and satisfaction with care; monthly utilization and costs; healthcare expenditure (out-of-pocket) and financing; and caregiver satisfaction / well being. There will be both unadjusted and adjusted measures. For time to first admission to nursing home, survival analysis specifically Cox Proportional Hazards regressions and intention-to-treat analysis will be carried out.

Since our study tracks participants over a period of 36 months, the first potential concern is participants in the control group who may be lost to follow-up 6 months after discharge which is when the MSW will close the care management files for patients. After the 6 months, the control group may for various reasons cease to receive community care unless they are in a VWO program that has care management. To minimize this difficulty, the available coordinated care management VWOs in the Bukit Merah catchment area will be provided with the list of names of the control group for oversight. Should any of the participants drop out of a community care program, the care coordinators can assist in enrolling the older adult in another care program should the participant decide that s / he would like to continue in a care program.

Statistical justification and the means by which data will be analyzed and interpreted

For the hypothesis to be tested, H03: Frail elderly in SingaPACE will have delayed first admission to institutionalized residential care nursing home relative to the frail elderly who are not in SingaPACE, survival analysis will be carried out. Shoenfeld's formula gives the total number of first nursing home admissions necessary to achieve 80% power as a function of the hazard ratio 32/(log HR)2. Assuming a hazard ratio of 0.35, along with first admission probabilities of 20% and 50% in SingaPACE and non-SingaPACE groups respectively, approximately 28 total admissions and therefore total participants (40 in each group) will be needed.

For the hypotheses H01: The elderly in SingaPACE will tend to have fewer admissions to accident & emergency (A&E) hospitalization than the elderly who are not in SingaPACE; H02: The elderly in SingaPACE will have fewer admissions to acute care hospitalization than the elderly who are not in SingaPACE; H04: The elderly in SingaPACE clients will have an enhanced QOL and satisfaction compared to the elderly who are not in SingaPACE; and H05: Caregivers of the elderly in SingaPACE will have a lower care-giving burden compared to caregivers of the elderly who are not in SingaPACE, Wilcoxon rank sum tests will be carried out. Assuming that observations from one group will exceed observations from the other group at least 55% of the time, each of these tests will have greater than 80% power for detecting a difference between the groups.

The analytical strategy will consist of hypothesis testing for each of the five individual hypotheses and intention-to-treat analysis. Also there will be an examination of the distributions of the main outcomes across all participants in each arm over 36 months. This will be complemented by a meta-analysis of the effectiveness of PACE programs in the US and Singapore.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 and above;
* The frail elderly classified as high Category2 - Category 3 under the Residence Assessment Form(RAF);
* Are willing to enroll in SingaPACE if they were selected in a fair lottery draw or to be followed up similarly over 36 months if not selected;
* Residing within the Bukit Merah catchment area;

Exclusion Criteria:

* Bed Bound;
* Are undergoing dialysis treatment,
* Radiotherapy or chemotherapy; or
* Have behavioral and psychological symptoms of dementia(BPSD)prior to enrollment in the research study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of EMT and acute care events | 36 months
  The primary outcome measure will be the number of EMT events, A&E visits or acute care hospitalizations captured based on the following possible sequence of events:
  * The number of EMT events or
  * The number of EMT events leading to A&E events or
  * The number of EMT events leading to A&E events that lead to acute care hospitalizations or
  * The number of A&E events or
  * The number of A&E events that lead to acute care hospitalizations or
  * The number of acute care hospitalizations

SECONDARY OUTCOMES:
Admission to institutionalized nursing home | 36 months
  From randomization point, time to first admission to nursing home over the 36 month period
Length of stay in acute care | 36 months
  For each acute care hospitalization, the length of stay
Patient Quality of Life | 36 months
  Patient QOL assessed using EQ-5D at 6 month intervals for the given time frame
Caregiver burden | 36 months
  Using the Zarit Caregiver Burden measure, assess changes to caregiver (spouse, family members, friends) burden at 6 month intervals for the given time frame

CONTACTS AND LOCATIONS:
Overall Officials: David B Matchar, MD,FACP,FAHA, Principal Investigator — Duke-NUS Graduate Medical School
Locations (2):
- Singapore (2):
  - NTUC Eldercare, Singapore
  - Tiong Bahru Central Plaza, Singapore